CLINICAL TRIAL: NCT03145415
Title: Comparison of Pudendal Nerve Block vs Caudal Block for Hypospadias Repair in Young Children: A Blinded Randomized Trial
Brief Title: Comparison of Pudendal Nerve Block and Caudal Block for Hypospadias in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: lh0001
Record Dates: First submitted 2017-05-03; First posted 2017-05-09 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2017-04

CONDITIONS: Hypospadias and Epispadias
Keywords: pudendal nerve block; hypospadias; caudal block
MeSH Terms: conditions — Hypospadias; Epispadias

STUDY DESIGN:
Intervention Model Description: All Children will be randomly assigned to one of 2 groups of 30 patients each using a computer generated number table.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: No other parties will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Pudendal block (Experimental): 0.25 cc per kg of 0.2% ropivacaine will be injected once for right pudendal N block and the same volume for the left pudendal N block before the start of the surgery
  Interventions: Procedure: Bilateral Pudendal block
- Caudal block (Active Comparator): 1 cc per kg of 0.2% ropivacaine in the caudal space given before the start of surgery
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Caudal block — 1 cc per kg of 0.2% ropivicaine in the caudal space given before the start of surgery.
  Arms: Caudal block
Procedure: Bilateral Pudendal block — 0.5 cc per kg of 0.2% ropivicaine. Half of the volume given as a right pudendal block and the remaining volume given on the left pudendal nerve block given prior to the start of surgery
  Arms: Bilateral Pudendal block

SUMMARY:
The purpose of this randomized blinded prospective study is to compare the analgesic efficacy and duration of a Pudendal Nerve Block (PNB) to a Caudal Block (CB) for pediatric patients, ages 6 months to 2 years, undergoing hypospadias repair.

DETAILED DESCRIPTION:
Hypospadias repair is one of the most common congenital malformations of the penis in the United States. It has an incidence of about 1 in 300 births. A combination of general anesthesia and a caudal block or general anesthesia combined with a pudendal nerve block are commonly used for hypospadias repair.

In our institution, hypospadias repair is typically done in infants and children ages 6 months to age two. A comparison of the efficacy of pudendal block versus the caudal block has not been undertaken in this younger population.

ELIGIBILITY:
Inclusion Criteria:

* Boys undergoing hypospadias repair

Exclusion Criteria:

-

Ages: 6 Months to 2 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | up to 24 hours
  The child's care giver will document the times that a rescue opioid was given to relieve pain.

SECONDARY OUTCOMES:
Intraoperative block assessment | up to 3 hours
  A heart rate increase above of 20 percent of baseline will be an indication of inadequate block that will be treated with a rescue opioid.
Post operative pain | up to 2 hours
  The FLACC scale scores greater than 6 will be an indication of inadequate pain relief needing a rescue dosages of opioid.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours/ duPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choudhry DK, Heredia L, Brenn BR, Brown M, Carvalho NF, Whaley MC, Shaik SS, Hagerty JA, Bani Hani A. Nerve stimulation guided bilateral pudendal nerve block versus landmark-based caudal block for hypospadias repair in young children: a prospective, randomized, pragmatic trial. Reg Anesth Pain Med. 2022 Dec;47(12):744-748. doi: 10.1136/rapm-2022-103680. Epub 2022 Sep 8. PMID 36283712